CLINICAL TRIAL: NCT06865196
Title: An Evaluation of Selected Teen Triple P as a Universal Intervention Delivered Through Telehealth
Brief Title: Investigating a Brief Virtual Seminar Series for Parents of Teens Ages 13-17
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: American Psychological Foundation (Other)
Responsible Party: Principal Investigator, John Cooley, Assistant Professor, University of Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-1035t
Record Dates: First submitted 2025-02-06; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Positive Parenting Skills
Keywords: Selected Teen Triple P; Parenting Intervention; Telehealth; Positive Parenting

STUDY DESIGN:
Intervention Model Description: Three study conditions compared: intervention-as-usual, intervention without an active discussion component, and waitlist control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention-as-usual (Experimental): 90-minute positive parenting seminars with active discussion component
  Interventions: Behavioral: Positive Parenting Seminar Series
- Intervention without an active discussion component (Experimental): 60-minute positive parenting seminars without an active discussion component
  Interventions: Behavioral: Positive Parenting Seminar Series
- Waitlist Control (No Intervention): Assessment-only waitlist control condition

INTERVENTIONS:
Behavioral: Positive Parenting Seminar Series — Selected Teen Triple P Positive Parenting Seminar Series Delivered Through Telehealth
  Other Names: Selected Teen Triple P
  Arms: Intervention without an active discussion component; Intervention-as-usual

SUMMARY:
The goal of this clinical trial is to see if a brief positive parenting seminar series delivered virtually helps parents of teenagers ages 13-17 learn additional tools and strategies to support teens' development, encourage good behavior, build confidence and responsibility, and improve how teens connect with others. The study also looks at how these seminars improve parenting practices and teen outcomes.

The main questions it aims to answer are whether parents are satisfied with the intervention and find the strategies helpful and acceptable, whether the intervention leads to changes in parenting behaviors (e.g., positive parenting) and teen outcomes (e.g., emotional and behavioral problems), and how removing the group discussion from the seminars impacts parents' ability to improve their parenting skills and their teenager's outcomes.

Researchers will compare three groups: parents receiving the seminars with a group discussion, parents receiving the seminars without a group discussion, and parents on a waitlist. This will help determine if group discussions lead to greater improvements in parenting practices and teen outcomes.

Participants will attend three online parenting seminars via telehealth (if assigned to a seminar group). They will complete surveys before, during, and after the seminars to share their experiences and provide feedback. Participants in the waitlist group will complete surveys at the beginning and end of the study, and will participate in the seminars after the study period.

DETAILED DESCRIPTION:
Despite the effectiveness of parenting interventions in promoting adaptive child-rearing behaviors and preventing youth internalizing and externalizing problems, our current model for mental health treatment that involves a highly trained mental health professional providing services in a one-on-one format at a clinic, private office, or health-care facility is not sustainable. As such, there is an urgent need to identify ways to increase the accessibility and scalability of mental health services to reduce the well-documented gap between youth and families who need mental health services and those who are able to access them. There is also a paucity of evidence-based parenting interventions for parents of adolescents, despite the increased risk for family conflict and mental health difficulties observed during this developmental period; thus, the primary goal of the current project is to examine the feasibility, acceptability, and preliminary efficacy of a brief (i.e., 3 session) seminar series for parents of adolescents between the ages of 13 and 17, which will be offered via telehealth to increase accessibility. Finally, this project will evaluate whether the ability for parents to ask questions and discuss skill implementation with a mental health provider is necessary for treatment effectiveness, given that programs that do not require a provider for implementation have the potential for greater scalability.

After completing the baseline survey, eligible parents will be randomly assigned to condition using block randomization. For parents assigned to the intervention-as-usual condition (i.e., 90-minute condition), seminars will be delivered live by two masters-level therapists who are fully accredited in Selected Teen Triple P. The seminars consist of 60-minutes of seminar content (i.e., discussion of various parenting strategies), followed by a 30-minute question-and-answer period. Participation will be encouraged by co-leaders throughout the seminars and the question-and-answer period.

For parents assigned to the intervention without an active discussion component (i.e., 60-minute condition), seminar content will be pre-recorded by the same two co-leaders who lead the seminars live to ensure standardization of the material and to create an environment focused on receiving information rather than active participation. During these meetings, participants will not be allowed to unmute and will only be able to message the hosts of the meeting (i.e., the leader).

The same seminar content was covered in both intervention conditions. The seminars included Raising Responsible Teenagers, Raising Competent Teenagers, and Getting Teenagers Connected.

Approximately 2-months and 4-months after attending the final seminar, parents will be contacted to complete a 30-minute follow-up survey for which they will be compensated. The dates that parents attended each seminar will be recorded and parents will be contacted approximately 2-months and 4-months after their last attended seminar (or their last opportunity to attend a seminar if they do not attend all three seminars). Parents in the waitlist control condition will be contacted approximately 2-months and 4-months after the last seminar was offered to those assigned to the intervention conditions in their enrollment cohort.

ELIGIBILITY:
Inclusion Criteria:

* Parent must reside in the State of Texas
* Parent has to have at least one child ages 13-17 years
* Teenager has to live with parent at least one night every 2 weeks

Exclusion Criteria:

* Parent does not have sufficient English proficiency to understand seminar content and complete study-related surveys
* Parent does not have access to the internet and/or can not attend seminars using the Zoom platform
* Teenager is currently participating in mental health services
* Teenager began taking psychiatric medication within 1 month of the study
* Parent is currently participating in mental health services

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Parent Satisfaction | Weekly, through intervention completion, average of 3 weeks.
  Parents assigned to an intervention condition will complete a modified 8-item version of the Parent Satisfaction Survey. Response options ranged from 1 (Poor, No definitely not, or Not at all) to 7 (Excellent, Yes, definitely, or Very much).
Acceptability | Weekly, through intervention completion, average of 3 weeks.
  Parents assigned to an intervention condition will complete a modified 9-item version of the Treatment Acceptability Rating Form. Response options range from 1 (Not at all) to 7 (Very much).
Positive Parenting | Baseline, 2-month, and 4-month follow-up assessments.
  All parents will complete the 16-item positive parenting composite measure of the Multidimensional Assessment of Parenting Scale, which is comprised of proactive parenting (6-items), positive reinforcement (4-items), warmth (3-items), and supportiveness (3-items) sub-scales. Response options range from 1 (Never) to 5 (Always) reflecting the frequency with which parents engage in different parenting behaviors.
Negative Parenting | Baseline, 2-month, and 4-month follow-up assessments.
  All parents will complete the 18-item negative parenting composite measure of the Multidimensional Assessment of Parenting Scale, which is comprised of hostility (7-items), physical control (4-items), and lax control (7-items) sub-scales. Response options range from 1 (Never) to 5 (Always) reflecting the frequency with which parents engage in different parenting behaviors.
Parental Psychological Control | Baseline, 2-month, and 4-month follow-up assessments.
  All parents will complete the 8-item Parent Psychological Control Measure, that is based off the Psychological Control Scale - Youth Self-Report. Response options range from 1 (Never) to 5 (Always) reflecting the frequency with which parents engage in different parenting behaviors.
Parental Monitoring | Baseline, 2-month, and 4-month follow-up assessments.
  All parents will complete the 9-item Parental Monitoring Scale and the 15-item Sources of Parental Knowledge scale. Responses range from 1 (No, never) to 5 (Yes, always), reflecting how often parents know information about their teenager's whereabouts and activities, and how they learn this information.
Parent-Adolescent Relationship | Baseline, 2-month, and 4-month follow-up assessments.
  All parents will complete the 4-item Involvement and 6-item Connectedness subscales of the Parent Adolescent Relationship Scale. Responses range from 0 (Not at all true) to 5 (Nearly always or always true) and reflect how true each statement was of parents' relationships with their teenager.
Parent-Teen Conflict | Baseline, 2-month, and 4-month follow-up assessments.
  All parents will complete a slightly modified version of the Aversive Parent-Child Interactions scale of the Youth Everyday Social Interactions and Mood measure. Responses range from 1 (Not at all) to 5 (A lot), reflecting the frequency with which there was conflict between parents and their teenager.
Parental Hope | Baseline, Weekly, through intervention completion (average of 3 weeks), 2-month, and 4-month follow-up assessments.
  All parents will complete the 5-item Hope for Parenting Scale. Response options range from 1 (Definitely False) to 8 (Definitely True) indicating how much they agree or disagree with each item.
Parental Self-Efficacy | Baseline, Weekly, through intervention completion (average of 3 weeks), 2-month, and 4-month follow-up assessments.
  All parents will complete the 5-item Brief Parental Self-Efficacy Scale. Response options range from 1 (Strongly Disagree) to 5 (Strongly Agree), indicating how much they agree with each statement.
Global Satisfaction | 2-month follow-up.
  Parents assigned to an intervention condition also completed the 8-item Client Satisfaction Questionnaire. Response options ranged from 1 (None of my needs have been met, Quite dissatisfied) to 4 (Almost all of my needs have been met, Very satisfied).

SECONDARY OUTCOMES:
Adolescent Emotional and Behavioral Difficulties | Baseline, 2-month, and 4-month follow-up assessments.
  All parents will complete the 25-item Strengths and Difficulties Questionnaire. This measure consists of emotional problems (5-items), conduct problems (5-items), hyperactivity (5-items), peer problems (5-items), and prosocial behavior (5-items) sub-scales. Each sub-scale will be examined as an outcome, along with the total difficulties scale, which is a composite of all five sub-scales and reflects overall emotional and behavioral difficulties. Response options range from 0 (Not true) to 2 (Certainly True) and reflects how often children experience various difficulties.
Adolescent Emotion Dysregulation | Baseline, 2-month, and 4-month follow-up assessments.
  All parents will complete the 24-item Emotion Dysregulation Inventory. Response options range from 0 (Not at all) to 4 (Very severe) reflecting the severity of various emotions and behaviors displayed by teenagers.
Adolescent Emotion Regulation | Baseline, 2-month, and 4-month follow-up assessments.
  All parents will complete the 8-item emotion regulation sub-scale of the Emotion Regulation Checklist. Response options range from 0 (Never) to 3 (Almost always) reflecting the frequency with which teenagers displayed various emotions and behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: John L. Cooley, Ph.D., Principal Investigator — University of Florida; Caroline Cummings, Ph.D., Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided